CLINICAL TRIAL: NCT04522492
Title: Impact of COVID-19 Pandemia on the Mental Health of Patients With Skin Picking Disorder and Their Treatment With Remote Cognitive Behavioral Therapy: Controlled Clinical Trial
Brief Title: Impact of COVID-19 on Mental Health of Patients With Skin Picking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 31520820.1.0000.5327
Record Dates: First submitted 2020-08-07; First posted 2020-08-21 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Skin Picking
MeSH Terms: conditions — Excoriation Disorder

STUDY DESIGN:
Intervention Model Description: randomized clinical trial with the intervention consisting of cognitive behavioral therapy in an online setting, and the control consisting of an active control group (guidelines about strategies to improve quality of life).
Who Masked: Outcomes Assessor
Masking Description: Two assessors will evaluate patients before and after the intervention, thru an online consultation and application of instruments to assess symptoms. The assessors will be blinded about the intervention received by the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- internet CBT (Experimental): Internet delivered cognitive behavioral therapy, thru 2 booster sessions. Each session will last 50 minutes. Fist session will involve: psychoeducation about the symptoms, evaluation of the skin picking habit, reinforcement of the habit reversal strategies. After 1 week, the second session will be applied, consisting of: strategies to cope with anxiety (breathing and muscle relaxation techniques) and to cope with depressive status (cognitive restructuring techniques).
  Interventions: Behavioral: Internet-based Cognitive Behavioral Therapy
- Quality of life promotion (Active Comparator): The therapist will send to the patient 2 videos with strategies to improve quality of life during the pandemia (1 video about social support and one video about sleep hygiene). After 1 week, the therapist will send to the patient another 2 videos with strategies do improve quality of life (dietary guidance and guidance on physical activity)
  Interventions: Other: Quality of life promotion

INTERVENTIONS:
Behavioral: Internet-based Cognitive Behavioral Therapy — 2 booster sessions of cognitive behavioral therapy (CBT) delivered thru internet to patients previously treated with CBT. First session focus on understanding the symptoms of skin picking and training techniques to reverse the habit. Second session focus on comorbid symptoms of anxiety and depression, training strategies to improve it.
  Arms: internet CBT
Other: Quality of life promotion — 2 videos about quality of life promotion will be send to patients in the active control arm. In the first week, the videos will consist in: social support techniques and sleep hygiene. After one week, 2 another videos will be send, consisting in: guide about healthy diet and about physical exercise.
  Arms: Quality of life promotion

SUMMARY:
Skin Picking Disorder (SPD) affects up to 10% of the general population, causing significant socioeconomic damage in 75% of affected individuals. It is characterized by the repeated habit of touching the skin itself, causing or aggravating wounds, with difficulty in controlling the habit. It is associated with anxiety disorders in about 20% of cases and with depressive disorder in about 50%. Patients with SPD have difficulties in regulating emotions, being more vulnerable to having their mental symptoms aggravated in face of stressful situations, such as the current coronavirus-19 pandemia. Among the treatments available to SPD, cognitive behavioral therapy is the only intervention superior to placebo, and there is still no medication approved by the FDA indicated specifically to SPD. The effectiveness of cognitive behavioral therapy was assessed in a randomized clinical trial with Brazilian patients with SPD, but its long-term benefit has not yet been evaluated. Additionally, telemedicine interventions can be effective and used during pandemia, but the effectiveness of internet delivered cognitive behavioral therapy for SPD is not clear yet.

DETAILED DESCRIPTION:
This study is a randomized clinical trial, in which patients diagnosed with skin picking disorder (SPD) will be evaluated and, if symptomatic for the disease, will be randomized to one of the arms: intervention arm with 2 booster sessions of cognitive behavioral therapy in online format; active control arm, in which individuals will watch videos with quality of life orientation. Patients included in this study are coming from a brazilian clinical trial conducted between the years of 2014 and 2018, in wich patients with SPD were treated with a cognitive behavioral treatment protocol in individual or group formats, resulting in improvement of SPD symptoms and comorbid anxiety and depression. Before the intervention, individuals will be evaluated by a psychiatrist, to assess SPD and comorbid symptoms severity, thru the application of some instruments to assess SPD, anxiety, depression and emotional regulation. Also, the CRISIS questionnaire, about the impact of COVID-19 in mental health, will be applied. After the interventions, the instruments will be applied again, by the same evaluator, wich is blinded to the type of intervention that the patient received.

ELIGIBILITY:
Inclusion Criteria:

* Skin picking as a primary diagnosis
* Treatment with cognitive behavioral therapy in the past, received in previous clinical randomized trial conducted by our research group between 2014 and 2018

Exclusion Criteria:

* Acute psychotic disorder, bipolar affective disorder in an acute episode, substance use disorder (except tobacco), severe depressive episode or suicidal ideation, dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Change in Global Clinical Impression Scale | 2 weeks
  The skin picking improvement after intervention will be assessed by the change in the Global Clinical Impression Scale, applied by blinded evaluators.

SECONDARY OUTCOMES:
Change in Beck Anxiety Inventory | 2 weeks
  Anxiety severity improvement after the intervention, assessed thru the Beck Anxiety Inventory
Change in Beck Depression Inventory | 2 weeks
  Depression severity improvement after the intervention, assessed thru the Beck Depression Inventory
Change of Skin Picking Impact Scale | 2 weeks
  Impact of Skin Picking in the life of the patient, assessed thru the Skin Picking Impact Scale
Change of emotional regulation | 2 weeks
  Assess the correlation of emotional regulation, thru the DERS-36 (difficulties in emotional regulation scale), with the different skin picking subtypes (focused or automatic), thru the Milwaukee scale of dermatillomania subtypes.
Change in Hamilton Anxiety Scale | 2 weeks
  Evaluate change in anxiety symptoms thru the Hamilton anxiety scale applied by blinded evaluators

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Blaya Dreher, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tucker BT, Woods DW, Flessner CA, Franklin SA, Franklin ME. The Skin Picking Impact Project: phenomenology, interference, and treatment utilization of pathological skin picking in a population-based sample. J Anxiety Disord. 2011 Jan;25(1):88-95. doi: 10.1016/j.janxdis.2010.08.007. Epub 2010 Aug 13. PMID 20810239
- [Background] Alexander JR, Houghton DC, Bauer CC, Lench HC, Woods DW. Emotion regulation deficits in persons with body-focused repetitive behavior disorders. J Affect Disord. 2018 Feb;227:463-470. doi: 10.1016/j.jad.2017.11.035. Epub 2017 Nov 10. PMID 29156359
- [Background] Torales J, O'Higgins M, Castaldelli-Maia JM, Ventriglio A. The outbreak of COVID-19 coronavirus and its impact on global mental health. Int J Soc Psychiatry. 2020 Jun;66(4):317-320. doi: 10.1177/0020764020915212. Epub 2020 Mar 31. PMID 32233719
- [Result] Xavier ACM, Souza CMB, Flores LHF, Prati C, Cassal C, Dreher CB. Improving skin picking diagnosis among Brazilians: validation of the Skin Picking Impact Scale and development of a photographic instrument. An Bras Dermatol. 2019 Sep-Oct;94(5):553-560. doi: 10.1016/j.abd.2018.10.001. Epub 2019 Sep 30. PMID 31777356
- [Result] Xavier ACM, de Souza CMB, Flores LHF, Bermudez MB, Silva RMF, de Oliveira AC, Dreher CB. Skin picking treatment with the Rothbaum cognitive behavioral therapy protocol: a randomized clinical trial. Braz J Psychiatry. 2020 Sep-Oct;42(5):510-518. doi: 10.1590/1516-4446-2019-0636. PMID 32401873